CLINICAL TRIAL: NCT01682265
Title: Stretta In Reflux Uncontrolled by Intake of Inhibitors of Protons Pump (IPP).- The SIRUP Trial- Multicentric, Randomized, Double Blind, Prospective Study
Brief Title: Stretta In Reflux Uncontrolled by IPP
Acronym: SIRUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BRD/11/06-Q
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stretta procedure (Experimental): Patient randomized in Stretta procedure arm will be hospitalized to have endoscopy and esophagus will receive radiofrequency.
  Control visits will then take place until Month 6. At this visit endoscopic control will take place.
  Interventions: Other: Stretta procedure
- Sham procedure (Sham Comparator): Patient randomized in Sham procedure arm will be hospitalized to have endoscopy. Material necessary to perform Stretta procedure will be inserted (like in Stretta procedure arm) BUT esophagus will not receive radiofrequency.
  Control visits will then take place until Month 6. At this visit endoscopic control will take place.
  Interventions: Other: Sham procedure

INTERVENTIONS:
Other: Stretta procedure
  Other Names: Radiofrequency of esophagus
  Arms: Stretta procedure
Other: Sham procedure — No radiofrequency delivered
  Arms: Sham procedure

SUMMARY:
The aim of the study is to compare the Stretta procedure and the Sham procedure efficiency 6months post-procedure in reflux uncontrolled by intake of Inhibitors of Protons Pump (IPP) patients.

DETAILED DESCRIPTION:
The study is over a period of 1 year. After checking eligibility, the patient will be randomised in double blind : stretta procedure /sham procedure. Control visits will take place after 4 weeks (on site), 8 weeks (by phone), 12 weeks (by phone), 18 weeks(on site) and 24 weeks(on site).During the 24 weeks visit, the therapeutic success will be evaluated.

In case of success, endoscopic control will be performed and the patient will come back on site at week 36 and 48 (end of study). In case of therapeutic failure, the stretta procedure will be proposed to the patient without breaking the blind for the 1st procedure. The procedure will be scheduled between week 24 and week 27. The patient will come back for a visit on site at weeks 31, 36 and 48 (end of visit)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* Severe or moderate heartburn (at least 3 heartburn times per week), persistent under treatment with IPP

Exclusion Criteria:

* Recent oeso-gastro-duodenal endoscopy(< 3 months)
* Oesophagitis > grade A
* Endobrachyoesophagus > C0M1
* Hiatal Hernia > 2 cm
* Symptoms insufficiently relieved with continued intake of IPP or with intake of IPP according to needs
* Predominant symptom of Gastrooesophageal reflux disease other than heartburn
* Patients contra-indicated for radiofrequency technique
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-03-26 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Efficiency of the treatment 6 months post-procedure | 6 months
  Evaluate the efficiency of the treatment 6 months post-procedure according to the patient's answers to the 2 following items : IPP treatment taken less than 7 days /week and adequate relief of symptoms. These results will be completed by the patient on a calendar during 2 weeks before the visit week 24

SECONDARY OUTCOMES:
Effects on digestive symptoms | 6 months
  Compare Stretta and sham procedure according to complete relief of digestive symptoms and pyrosis (calculation based upon number of days without digestive symptoms and pyrosis as indicated by the patient on a questionary completed during the 2 weeks preceding visits à 6 months)
Effects on digestive symptoms | 1 year
  Compare Stretta and sham procedure according to complete relief of digestive symptoms and pyrosis (calculation based upon number of days without digestive symptoms and pyrosis as indicated by the patient on a questionary completed during the 2 weeks preceding visits à 12 months)
Necessity of IPP treatment | 6 months
  Compare Stretta and sham procedure according to necessity of IPP treatment
necessity of IPP treatment | 1 year
  Compare Stretta and sham procedure according to necessity of IPP treatment
Tolerance | 6 months
  Compare Stretta and sham procedure according to Tolerance analysed by recording of adverse events (sides effects of each procedure) until week 24.
Tolerance | 1 year
  Compare Stretta and sham procedure according to Tolerance analysed by recording of adverse events (sides effects of each procedure) until week 48.
Quality of live | 6 months
  Compare Stretta and sham procedure according to Quality of life (use of quality of life questionaries)
Quality of life | 1 year
  Compare Stretta and sham procedure according to Quality of life
pH-impedancemetry predictive factors | At Inclusion
  pH-impedancemetry will be realized at clinical trial start, when patient is under PPI intake to determine pH-impedancemetry predictive factors for positive response to stretta method. Acid and non acid exposition of the esophagus will be measured as well as the SAP (Symptom Association Probability) which corresponds to the probability of association between symptoms felt by the patient during the pH-impedancemetry and episodes of acid or non acid reflux.
Efficiency | 1 year
  Evaluate efficiency of the stretta procedure in patients unsatisfied after the sham procedure at week 48 according to the patient's answers to the 2 following items : IPP treatment taken less than 7 days /week and adequate relief of symptoms. These results will be completed by the patient on a calendar during 2 weeks before the visit week 48
Efficiency | 1 year
  Evaluate efficiency of the 2nd stretta procedure in patients unsatisfied after the 1st stretta procedure at week 48 according to the patient's answers to the 2 following items : IPP treatment taken less than 7 days /week and adequate relief of symptoms. These results will be completed by the patient on a calendar during 2 weeks before the visit week 48

CONTACTS AND LOCATIONS:
Overall Officials: Stanislas Bruley des Varannes, Professor, Principal Investigator — Nantes Universitary Hospital; Chloe Melchior, Doctor, Principal Investigator — Rouen Universitary Hospital; Thierry Ponchon, Professor, Principal Investigator — Lyon Universitary Hospital; Franck Zerbib, Professor, Principal Investigator — Bordeaux Universitary Hospital; Franck Cholet, Doctor, Principal Investigator — Brest Universitary hospital; Benoit Coffin, Professor, Principal Investigator — APHP-Louis Mourier hospital
Locations (6):
- France (6):
  - Nantes Universitary Hospital, Nantes, Loire Atlantique
  - Bordeaux Universitary Hospital, Bordeaux
  - Brest universitary hospital, Brest
  - APHP - Louis Mourier hospital, Colombes
  - Lyon Universitary Hospital, Lyon
  - Rouen Universitary Hospital, Rouen

REFERENCES:
- [Derived] Zerbib F, Sacher-Huvelin S, Coron E, Coffin B, Melchior C, Ponchon T, Cholet F, Chabrun E, Vavasseur F, Gorbatchef C, Zalar A, Mion F, Robaszkiewicz M, Le Rhun M, Leroy M, Paul Galmiche J, Bruley des Varannes S. Randomised clinical trial: oesophageal radiofrequency energy delivery versus sham for PPI-refractory heartburn. Aliment Pharmacol Ther. 2020 Aug;52(4):637-645. doi: 10.1111/apt.15936. Epub 2020 Jul 13. PMID 32656869